CLINICAL TRIAL: NCT06186661
Title: The Effect of Cognitive Rehabilitation Based on Multicontextual Treatment Approach in Stroke: A Randomized Controlled Trial
Brief Title: Multicontextual Treatment Approach in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ozden erkan (Other)
Collaborators: Florence Nightingale Hospital, Istanbul (Other); Memorial Sisli Hospital, Istanbul (Other)
Responsible Party: Sponsor-Investigator, ozden erkan, assistant professor, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410-01-3346
Record Dates: First submitted 2022-09-02; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Stroke; Cognitive Impairment; Quality of Life
Keywords: social participation; occupational therapy; stroke; cognition; quality of life
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Experimental group was applied a total of 2 hours-exercise programs consisting of 1-hour-neurophysiological exercise and 1-hour cognitive rehabilitation
  Interventions: Other: neurophysiological exercise; Other: cognitive rehabilitation
- Control Group (Active Comparator): The Control Group was implemented only 1-hour neuropsychological exercise program.
  Interventions: Other: neurophysiological exercise

INTERVENTIONS:
Other: neurophysiological exercise — The content of the treatment program consisted of neurophysiological exercises based on Bobath.
Other: cognitive rehabilitation — Cognitive rehabilitation sessions of the experimental group included 30 minutes of remedial and functional adaptive approaches and 30 minutes of implementation of Multicontextual treatment intervention.
  Arms: Experimental Group

SUMMARY:
BACKGROUND: It is known that cognitive disorders affect the rehabilitation of stroke patients but which cognitive rehabilitation intervention should apply to stroke patients and what their effects are on their life is not clear yet.

OBJECTIVE: to investigate the effects of cognitive rehabilitation including combined approaches on quality of the life and social participation of stroke patients.

METHODS: 20 patients with chronic stroke were randomly divided into two groups (Group 1 and 2), each including 10. Patients in each group were treated with neurophysiological exercises 3 times a week for 8 weeks and the subjects in Group 1 received cognitive rehabilitation additionally. The cognitive rehabilitation program consisted of individualized combined approaches including multicontextual treatment and bottom-up approaches. Loeweinstein Occupational Therapy Cognitive Assessment (LOTCA), Montreal Cognitive Assessment (MoCA) to assess cognitive status, Short Form-36 (SF-36) to assess the quality of life, Functional Independence Measure (FIM) to evaluate functional independence, Canadian Occupational Performance Measure and Craig Handicap Assessment and Reporting Technique- Short Form (CHART-SF) to evaluate social participation were used.

DETAILED DESCRIPTION:
Forty-two patients who were diagnosed with a stroke by a neurologist were admitted to the Stroke Unit of Sisli Memorial Hospital from November 2011 to April 2014. Our study was conducted on 20 patients who met the inclusion criteria of the study. Informed consent was obtained from each patient before the study. The Ethics Commission of Hacettepe University Senate (application No: 410.01-3346) approved this study. Patients were randomly divided into two groups of 10 people using a random number table. The number of cases was determined to be 10 patients for each group by using the power analysis method. Power analysis was performed based on the LOTCA and MoCA scales which are expected to have the most changes after the therapy. In this small randomized controlled trial (Small RCT); while the first group (CRG) applied a neurophysiological and cognitive rehabilitation therapy consisting of individualized combined approaches including multi-contextual treatment and bottom-up approaches, the second group (CG) implemented only a neurophysiological treatment program as the control group.

The 1st group determined by randomization applied a total of 2 hours-exercise programs consisting of 1-hour-neurophysiological exercise and 1-hour cognitive rehabilitation. The 2nd Group implemented only a 1-hour neuropsychological exercise program. The treatment programs determined for both groups were carried out 3 days a week for a total of 8 weeks. Cognitive rehabilitation sessions of the 1st group included 30 minutes of remedial and functional adaptive approaches and 30 minutes of implementation of Multicontextual treatment intervention.

While determining the cognitive rehabilitation programs of the patients; the weak areas in their cognitive skills were identified by analyzing the tests conducted before the treatment. Restorative approaches consisted of the repetition of pencil-and-paper activities and computer-based exercises according to the weak cognitive skills of the patients determined by the assessments made.

While determining a specific multi-contextual treatment intervention for the patients; their roles, personalities, habits, interests, requests, living conditions, and environments were questioned, the activities determined by COPM were revised and the essential requirements of this approach tried to be ensured.

According to this approach, using multiple environments and conditions, transfer of learning, and increasing the patient's awareness were provided. Also, the usage of various strategies and associating the new knowledge with the old knowledge were emphasized

ELIGIBILITY:
Inclusion Criteria:

* Patients with the first time diagnosis of stroke, between 18-80 age range, a post-stroke period of a minimum of 6 and maximum of 24 months, with 21 or less scores on the Montreal Cognitive Assessment Scale(MoCA), who gained the sitting and standing balance and who were able to communicate enough to understand simple orders were included in the study

Exclusion Criteria:

* with pre-stroke dementia or Alzheimer's diagnosis, who had vision problems and developed post-stroke aphasia, were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07-04 (Actual); Primary Completion 2011-08-29 (Actual); Study Completion 2014-06-13 (Actual)

PRIMARY OUTCOMES:
Change outcome measure: Montreal Cognitive Assessment | pre-treatment and 8 weeks
  It has been developed to assess mild cognitive impairments, assesses several cognitive domains; executive functions, visuo-constructional skills, memory, language, attention and concentration, conceptual thinking, calculations, and orientation
Change outcome measure: Loewenstein Occupational Therapy Cognitive Assessment | pre-treatment and 8 weeks
  It has been developed to assess the basic cognitive skills in individuals with a brain damage that is caused by traumatic head injuries, stroke, and brain tumors.The LOTCA scale, the validity of which has been proved by the conducted studies so far, consists of a total of 26 subtests within 6 main areas: orientation, visual perception, spatial perception, motor praxis, visuomotor organization, and thinking operations. A high score indicates complete cognitive skills.
Change outcome measure: Canadian Occupational Performance Measure (COPM) | pre-treatment and 8 weeks
  The COPM is a reliable and valid semi-structured interview measurement tool. Its reliability and validity in the patient groups with stroke have been proved.A high score indicates high performance and satisfaction.

SECONDARY OUTCOMES:
Change outcome measure: Craig HandicapAssessment and Reporting Technique-Short Form-(CHART-SF) | pre-treatment and 8 weeks
  It has developed to determine individuals' level of disability in their social lives, is isused for various populations such as stroke, spinal cord injury, traumatic brain injury, and multiple sclerosis. The maximum score of 100 represents the level of participation of the person without a disability.
Change outcome measure: Functional Independence Measure (FIM) | pre-treatment and 8 weeks
  Consisting of 18 items, the FIM has two main sections that evaluate motor (13 items) and cognitive functions (5 items). These two main sections are also evaluated with subgroups within themselves. A high score indicates complete independence.

CONTACTS AND LOCATIONS:
Overall Officials: Özden E OGUL, PhD, Principal Investigator — Medipol University; Gonca BUMIN, PhD, Study Chair — Hacettepe University; Yakup KRESPİ, MD, Study Director — Istınye University /Istanbul
Locations (1):
- Florence Nightingale Hospital Stroke Center and Şişli Memorial Hospital, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No